CLINICAL TRIAL: NCT01860300
Title: Multicentre, Randomised, Double-blinded, Placebo-controlled Trial of Efficacy of Amoxicilline/Clavulanic Acid in Patients Affected by Tic Disorder Colonized by Group A Streptococcus
Brief Title: Efficacy of Amoxicilline/Clavulanic Acid in Patients Affected by Tic Disorder Colonized by Group A Streptococcus
Acronym: AntibioTICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Cardona, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sapienza Università di Roma; 2012-002430-36 (EudraCT Number)
Record Dates: First submitted 2013-05-19; First posted 2013-05-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Tic Disorders
Keywords: Tic Disorders; Tourette Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic (Experimental): Amoxicillin-Potassium Clavulanate Combination
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate Combination — Amoxicillin-Potassium Clavulanate Combination will be prescribed at the dose of 25/3.6 mg/kg/day for 10 days, 2 times/day, as oral suspension.
  Other Names: Augmentin
  Arms: Antibiotic
Drug: placebo
  Arms: Placebo

SUMMARY:
This study is an extension of the European Multicentre Tics In Children Studies (EMTICS) COURSE study for which a separate study protocol exists; Aim of this clinical trial is to study the efficacy of treatment with antibiotics in reducing severity of tics and associated neuropsychiatric symptoms in patients with a tic disorder colonised by GAS.

Primary Objective: Test the hypothesis that antibiotic treatment of GAS colonisation compared to placebo is associated with a larger reduction of tic and associated neuropsychiatric symptoms in the short-term (1 month) in patients with a tic disorder colonised by GAS.

Secondary Objective: Test the hypothesis that antibiotic treatment of GAS colonisation is superior to placebo in the long-term (1 year) reduction of tic and associated neuropsychiatric symptoms in patients with a tic disorder colonized by GAS.

Patients affected by a chronic tic disorder followed in the EMTICS- Longitudinal Course Study that show a positive culture for GAS at any microbiological examination during their follow-up will be considered eligible for the treatment trial.

Patients showing GAS positivity will be invited to participate in the clinical trial.

The patients enrolled will be randomly assigned to antibiotic or placebo in a 1:1 ratio.

All participating patients will undergo a microbiological, serological and clinical assessment 1 month after the date of entering in the treatment trial (i.e. around 20 days after the end of treatment). Then, the patients will be followed with clinical, laboratory and microbiological assessments every four months for 1 year.

Patients will be deblinded at the end of the treatment trial follow-up (1 year after the recruitment).

Patients who will develop a true GAS infection or who otherwise need to be prescribed antibiotics for any clinical reason during the follow-up will be withdrawn from the study and immediately deblinded. Data of such patients would, however, remain part of the study analyses, following the intention-to-treat principle.

DETAILED DESCRIPTION:
Following the few studies performed on this topic, children affected by tic disorder show a rate of Group A Streptococcus (GAS) colonization similar or slightly higher than that reported in the normal population.

However, several studies have documented high rates of elevated anti-streptolysin O titers (ASOT) in children affected by tic disorders. One study reported a significantly higher ASOT in 150 children with tics compared to 150 healthy children, documenting a direct relationship between ASOT and tic severity. In this study, however, throat swab culture analyses on a subsample of patients failed to detect a predominant GAS serotype associated with tics. An American cohort of 81 patients with TS also exhibited higher ASOT than age-matched healthy volunteers and a mixed group of patients with autoimmune diseases. Increased ASOT, anti-deoxyribonuclease B (DNAse B), anti- streptococcal M12 and M19 titres were also observed in a smaller German sample of patients with TS. In a British cohort of 100 patients with TS (50% children), ASOT was raised in 64% of children and in 68% of adults with TS; this was significantly higher than in neurological disease and healthy control subjects. Two other reports from British and Italian cohorts confirmed these findings. However, a subsequent study failed to find a significant association with ASOT and anti-DNAse B titres using the same cross-sectional approach. More recently, a study on a large service-based cohort of TS patients confirmed the significant elevated rate of the high ASOT, but evidenced also that, on prospective analysis, ASOT were persistently elevated in 57% of patients with TS. Moreover, in tic patients the enhanced immune response is not limited to ASOT but it involves a broad range of GAS antigens.

Taken together, these observations lead to hypothesize that TS patients colonized by GAS are not merely carriers and that this colonization may promote a sustained anti-streptococcal immune response contributing to the persistence of tic symptoms.

If this hypothesis is true, the antibiotic treatment of GAS colonization in patients affected by a chronic tic disorder could modify their symptoms in term of severity and number of exacerbations.

Up to now, only tic patients diagnosed as Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infection (PANDAS) underwent a controlled antibiotic treatment: two trials, aimed to study the efficacy of different preventive regimens on number of tic exacerbations, obtained however mixed results, mainly due to poor compliance.

Investigators here designed a placebo-controlled trial with amoxicilline/clavulanic acid in tic patients showing GAS colonization. This drug is the first line therapy for streptococcal pharyngo-tonsillitis. Some previous studies have shown a superiority of amoxicillin versus penicillin in the treatment of GAS infections. A 10-day course of amoxicillin is considered sufficient and efficient in the treatment of GAS tonsillo-pharyngitis. Moreover, oral amoxicillin/clavulanic acid and oral clindamycin for 10 days achieved comparable rates of bacteriologic eradication at 12 days and 3 months. Furthermore, amoxicilline/clavulanic acid has been demonstrated to be efficacious in the treatment of GAS colonization. A few antibiotic regimens - evaluated prospectively in randomized, controlled trials- have demonstrated efficacy for termination of GAS carriage: among these, a regimen of 10 days of amoxicillin/ clavulanic acid was more effective than repeat penicillin in patients with treatment failure. Thus, the 10-days regimen of amoxicilline/clavulanic acid should be efficient in GAS eradication and, on the other hand, the shortness of the treatment should avert problems in patient's compliance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tourette Syndrome or another chronic tic disorder according to DSM IV-TR criteria.
* Evidence of GAS colonization at any visit of EMTICS Longitudinal Course Study.
* Either no current psychotropic medication or on stable anti-tic medication for at least 2 months before the enrolment in the trial.
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Children and/or parents are unable to understand and comply with protocol
* Any antibiotic treatment for any reason during the last month before enrolment in the trial.
* Clinical manifestations of pharyngitis or other streptococcal infections at moment of enrolment in the trial.
* Known or suspected hypersensitivity to penicillin or other β-lactam antibacterials, a history of amoxicillin-clavulanate-associated cholestatic jaundice or hepatic dysfunction.
* Known and/or suspected renal or hepatic impairment (due to the potential for drug-related toxicity in patients with such a condition).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Severity of tic disorder | one month
  YGTSS scores

SECONDARY OUTCOMES:
Severity of tic disorder | one year
  YGTSS scores

OTHER OUTCOMES:
Severity of associated neuropsychiatric symptoms | one month - one year
  CYBOCS - PUTS - SCQ - SNAP-IV -SDQ

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cardona, MD, Principal Investigator — Sapienza Università di Roma
Locations (1):
- Department of Pediatrics and Child Neuropsychiatry, Rome, Italy

REFERENCES:
- [Background] Bombaci M, Grifantini R, Mora M, Reguzzi V, Petracca R, Meoni E, Balloni S, Zingaretti C, Falugi F, Manetti AG, Margarit I, Musser JM, Cardona F, Orefici G, Grandi G, Bensi G. Protein array profiling of tic patient sera reveals a broad range and enhanced immune response against Group A Streptococcus antigens. PLoS One. 2009 Jul 22;4(7):e6332. doi: 10.1371/journal.pone.0006332. PMID 19623252
- [Background] Cardona F, Orefici G. Group A streptococcal infections and tic disorders in an Italian pediatric population. J Pediatr. 2001 Jan;138(1):71-5. doi: 10.1067/mpd.2001.110325. PMID 11148515
- [Background] Church AJ, Dale RC, Lees AJ, Giovannoni G, Robertson MM. Tourette's syndrome: a cross sectional study to examine the PANDAS hypothesis. J Neurol Neurosurg Psychiatry. 2003 May;74(5):602-7. doi: 10.1136/jnnp.74.5.602. PMID 12700302
- [Background] Creti R, Cardona F, Pataracchia M, Hunolstein CV, Cundari G, Romano A, Orefici G. Characterisation of group A streptococcal (GAS) isolates from children with tic disorders. Indian J Med Res. 2004 May;119 Suppl:174-8. PMID 15232189
- [Background] Curtin-Wirt C, Casey JR, Murray PC, Cleary CT, Hoeger WJ, Marsocci SM, Murphy ML, Francis AB, Pichichero ME. Efficacy of penicillin vs. amoxicillin in children with group A beta hemolytic streptococcal tonsillopharyngitis. Clin Pediatr (Phila). 2003 Apr;42(3):219-25. doi: 10.1177/000992280304200305. PMID 12739920
- [Background] Garvey MA, Perlmutter SJ, Allen AJ, Hamburger S, Lougee L, Leonard HL, Witowski ME, Dubbert B, Swedo SE. A pilot study of penicillin prophylaxis for neuropsychiatric exacerbations triggered by streptococcal infections. Biol Psychiatry. 1999 Jun 15;45(12):1564-71. doi: 10.1016/s0006-3223(99)00020-7. PMID 10376116
- [Background] Kaplan EL, Johnson DR. Eradication of group A streptococci from the upper respiratory tract by amoxicillin with clavulanate after oral penicillin V treatment failure. J Pediatr. 1988 Aug;113(2):400-3. doi: 10.1016/s0022-3476(88)80291-9. No abstract available. PMID 3135377
- [Background] Loiselle CR, Wendlandt JT, Rohde CA, Singer HS. Antistreptococcal, neuronal, and nuclear antibodies in Tourette syndrome. Pediatr Neurol. 2003 Feb;28(2):119-25. doi: 10.1016/s0887-8994(02)00507-6. PMID 12699862
- [Background] Mahakit P, Vicente JG, Butt DI, Angeli G, Bansal S, Zambrano D. Oral clindamycin 300 mg BID compared with oral amoxicillin/clavulanic acid 1 g BID in the outpatient treatment of acute recurrent pharyngotonsillitis caused by group a beta-hemolytic streptococci: an international, multicenter, randomized, investigator-blinded, prospective trial in patients between the ages of 12 and 60 years. Clin Ther. 2006 Jan;28(1):99-109. doi: 10.1016/j.clinthera.2006.01.006. PMID 16490583
- [Background] Martino D, Church AJ, Defazio G, Dale RC, Quinn NP, Robertson MM, Livrea P, Orth M, Giovannoni G. Soluble adhesion molecules in Gilles de la Tourette's syndrome. J Neurol Sci. 2005 Jul 15;234(1-2):79-85. doi: 10.1016/j.jns.2005.03.032. PMID 15941572
- [Background] Martino D, Chiarotti F, Buttiglione M, Cardona F, Creti R, Nardocci N, Orefici G, Veneselli E, Rizzo R; Italian Tourette Syndrome Study Group. The relationship between group A streptococcal infections and Tourette syndrome: a study on a large service-based cohort. Dev Med Child Neurol. 2011 Oct;53(10):951-7. doi: 10.1111/j.1469-8749.2011.04018.x. Epub 2011 Jun 17. PMID 21679362
- [Background] Morshed SA, Parveen S, Leckman JF, Mercadante MT, Bittencourt Kiss MH, Miguel EC, Arman A, Yazgan Y, Fujii T, Paul S, Peterson BS, Zhang H, King RA, Scahill L, Lombroso PJ. Antibodies against neural, nuclear, cytoskeletal, and streptococcal epitopes in children and adults with Tourette's syndrome, Sydenham's chorea, and autoimmune disorders. Biol Psychiatry. 2001 Oct 15;50(8):566-77. doi: 10.1016/s0006-3223(01)01096-4. PMID 11690591
- [Background] Muller N, Kroll B, Schwarz MJ, Riedel M, Straube A, Lutticken R, Reinert RR, Reineke T, Kuhnemund O. Increased titers of antibodies against streptococcal M12 and M19 proteins in patients with Tourette's syndrome. Psychiatry Res. 2001 Mar 25;101(2):187-93. doi: 10.1016/s0165-1781(01)00215-3. PMID 11286821
- [Background] Rizzo R, Gulisano M, Pavone P, Fogliani F, Robertson MM. Increased antistreptococcal antibody titers and anti-basal ganglia antibodies in patients with Tourette syndrome: controlled cross-sectional study. J Child Neurol. 2006 Sep;21(9):747-53. doi: 10.1177/08830738060210091001. PMID 16970879
- [Background] Snider LA, Lougee L, Slattery M, Grant P, Swedo SE. Antibiotic prophylaxis with azithromycin or penicillin for childhood-onset neuropsychiatric disorders. Biol Psychiatry. 2005 Apr 1;57(7):788-92. doi: 10.1016/j.biopsych.2004.12.035. PMID 15820236